CLINICAL TRIAL: NCT05030285
Title: Telehealth Psychotherapy for Anxiety in Persons With Cognitive Impairment
Acronym: Tele-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC/17/QRBW/676
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Psychotherapy; Cognitive Impairment; Anxiety
Keywords: Psychotherapy; Cognitive Impairments; Anxiety
MeSH Terms: conditions — Cognitive Dysfunction; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomised (1:1 ratio) to either the Tele-CBT intervention or usual care (Control) arm.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded to what arm the participant is allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): People who are randomised into the intervention arm will undergo 6 weekly psychotherapy sessions
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Control (No Intervention): People who are randomised into the control arm will undergo usual care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — The CBT intervention includes 6 sessions via video-conferencing that has been tailored for people living with cognitive impairment. The sessions incorporate the use of psychoeducation and relaxation videos to improve home-based practise for long-term outcomes.
  Arms: Intervention

SUMMARY:
This project will pilot a tailored Cognitive Behavioral Therapy (CBT) intervention delivered via telehealth videoconferencing (Tele-CBT) to reduce anxiety in people living with cognitive impairment. A process evaluation will inform its feasibility and implementation in the community nation-wide.

DETAILED DESCRIPTION:
Anxiety is a pre-existing mental health issue in older persons with cognitive impairment (includes people with mild cognitive impairment (MCI) and dementia), with considerably high prevalence (14%) as compared to older persons in the general population (3%). Anxiety results in accelerated cognitive decline, increased aggressive behaviours, and even an increased risk of suicide. Anxiety also negatively influences quality of life (QoL) of the individual with cognitive impairment and their care partner, increases early institutionalisation, and amplifies economic burden.

The Tele-CBT package used in this study is a modification of existing manualised psychotherapeutic interventions for treatment of anxiety in people with Parkinson's disease and older adults with cognitive impairment. This new package incorporates techniques tailored to reduce anxiety in people with cognitive impairment, including symptom monitoring. The interventions will include various psychological techniques aimed at reducing anxiety and stress. The intervention consists of 6 weekly psychotherapy sessions. Each therapy session lasts between 30-60 minutes, depending on the participants' capacity to actively participate in session and on their cognitive functioning (e.g. complex attention, executive function). Support persons will be invited and instructed to actively engage in the therapy sessions as well as in between-session home tasks to support the person with cognitive impairment. These techniques will be facilitated via the use of non-immersive videos in telehealth videoconferencing.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a diagnosis of mild cognitive impairment (MCI) or dementia of any aetiology based on a previous diagnosis by a clinician or scoring above threshold (≤32; MCI ≤32 and dementia ≤27) for cognitive impairment in the Modified Telephone Interview for Cognitive Impairment (TICS-M).
* Persons screening positive for anxiety (scoring ≥9 in the Geriatric Anxiety Inventory, GAI) or reports subjective complaints of anxiety

Exclusion Criteria:

* Persons with severe dementia
* Persons who are unable to communicate or complete questionnaires
* Persons who are at high risk of suicide as identified by by the University of Queensland Suicidal Risk Assessment administered at the UQ Psychology clinic which has been modified for use by the Dementia and Neuro Mental Health Research Unit
* Persons who have major depression as the primary complaint without reported symptoms of anxiety.
* Persons on existing anxiolytics or antidepressants who have not been on a stable dose for at least 12 weeks before starting the trial and are unable to maintain the same dose for the duration of the trial. Changes to medication will be checked at each therapy and assessment session.
* Persons who are undergoing psychological therapy or will undergo psychological therapy over the trial duration.

Entry into the study:

Study entry will be determined by discussions with the core investigator team consisting of clinicians and experienced researchers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-07-16 (Actual); Study Completion 2022-07-16 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | Post assessment (week 8). Scores ranging between 0 to 54 (lower score indicates better outcomes)
  Change from baseline in anxiety as measured by the Rating Anxiety in Dementia Scale (RAID).

SECONDARY OUTCOMES:
Change in depression | Post assessment (week 8). Scores ranging between 0 to 15 (lower score indicates better outcomes)
  Change from baseline in depression as measured by the Geriatric Depression Scale (GDS)
Change in quality of life | Post assessment (week 8). Scores ranging between 0 to 52 (higher score indicates better outcomes)
  Change from baseline in quality of life as measured by the Quality of Life in Alzheimer's Disease (QoL-AD)
Change in carer burden | Post assessment (week 8). Scores ranging between 0-88 (lower score indicates better outcomes)
  Change from baseline in carer burden as measured by the Zarit Burden Inventory (ZBI)

CONTACTS AND LOCATIONS:
Overall Officials: Nadeeka Dissanayaka, PhD, Principal Investigator — The University of Queensland
Locations (1):
- The University of Queensland, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Kuring JK, Mathias JL, Ward L. Prevalence of Depression, Anxiety and PTSD in People with Dementia: a Systematic Review and Meta-Analysis. Neuropsychol Rev. 2018 Dec;28(4):393-416. doi: 10.1007/s11065-018-9396-2. Epub 2018 Dec 7. PMID 30536144
- [Background] Banks SJ, Raman R, He F, Salmon DP, Ferris S, Aisen P, Cummings J. The Alzheimer's disease cooperative study prevention instrument project: longitudinal outcome of behavioral measures as predictors of cognitive decline. Dement Geriatr Cogn Dis Extra. 2014 Dec 18;4(3):509-16. doi: 10.1159/000357775. eCollection 2014 Sep-Dec. PMID 25685141
- [Background] Ferretti L, McCurry SM, Logsdon R, Gibbons L, Teri L. Anxiety and Alzheimer's disease. J Geriatr Psychiatry Neurol. 2001 Spring;14(1):52-8. doi: 10.1177/089198870101400111. PMID 11281317
- [Background] Seyfried LS, Kales HC, Ignacio RV, Conwell Y, Valenstein M. Predictors of suicide in patients with dementia. Alzheimers Dement. 2011 Nov;7(6):567-73. doi: 10.1016/j.jalz.2011.01.006. PMID 22055973
- [Background] Poon E. A Systematic Review and Meta-Analysis of Dyadic Psychological Interventions for BPSD, Quality of Life and/or Caregiver Burden in Dementia or MCI. Clin Gerontol. 2022 Jul-Sep;45(4):777-797. doi: 10.1080/07317115.2019.1694117. Epub 2019 Nov 22. PMID 31752633
- [Background] Konnopka A, Konig H. Economic Burden of Anxiety Disorders: A Systematic Review and Meta-Analysis. Pharmacoeconomics. 2020 Jan;38(1):25-37. doi: 10.1007/s40273-019-00849-7. PMID 31646432